CLINICAL TRIAL: NCT07267247
Title: Cancer Therapy-Related Cardiac Dysfunction Associated With EGFR-TKIs in Advanced EGFR-mutant Non-small Cell Lung Cancer: A Single-center Prospective Observational Study
Brief Title: Cancer Therapy-Related Cardiac Dysfunction Associated With EGFR-TKIs in Advanced EGFR-mutant Non-small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Mu Han, Peng, Attending Physician, Department of Chest Medicine, Taichung Veterans General Hospital, Taichung Veterans General Hospital
Other Study IDs: VGHTC-CM-MHP-20250918
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer (MeSH Term: Carcinoma, Non-Small-Cell Lung); Drug-Related Side Effects and Adverse Reactions (MeSH Term); Egfr Tyrosine Kinase Inhibitor; Cardiotoxicity
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cardiotoxicity | interventions — EGFR tyrosine kinase inhibitor 324674

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: EGFR-TKI — Erlotinib, dacomitinib, afatinib, and osimertinib, with dose according to NCCN guide line.
Other: EGFR tyrosine kinase inhibitor — Erlotinib, dacomitinib, afatinib, and osimertinib, with dose according to NCCN guide line

SUMMARY:
This study investigated the incidence of cardiac dysfunction in patients with advanced or recurrent epidermal growth factor receptor (EGFR)-mutant non-small cell lung cancer treated with EGFR- tyrosine kinase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* patients with advanced or recurrent EGFR-mutant NSCLC receiving EGFR-TKI treatment

Exclusion Criteria:

* NIL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) with advanced or metastatic non-small cell lung cancer (NSCLC) harboring EGFR mutations, who are prescribed EGFR tyrosine kinase inhibitors (gefitinib, erlotinib, afatinib, dacomitinib, or osimertinib) as part of routine clinical care at Taichung Veterans General Hospital. All participants will undergo echocardiographic assessment at baseline and follow-up time points according to the study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
The incidence of cancer therapy-related cardiac dysfunction after treatment with EGFR tyrosine kinase inhibitors. | From enrollment to 2 years after initiating EGFR tyrosine kinase inhibitor treatment.
  Cancer therapy-related cardiac dysfunction was defined as a left ventricular ejection fraction of less than 50% and an absolute reduction in LVEF of more than 10% from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided